CLINICAL TRIAL: NCT01384175
Title: Epidural Anesthesia and Postoperative Analgesia With Ropivacaine and Fentanyl in Off-pump Coronary Artery Bypass Grafting
Brief Title: Epidural Anesthesia and Postoperative Analgesia With Ropivacaine and Fentanyl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Mikhail Kirov, Professor, Northern State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPCAB-EA
Record Dates: First submitted 2011-06-17; First posted 2011-06-28 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Artery Disease
Keywords: Epidural Analgesia; OPCAB; PCEA
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- intravenous analgesia (Active Comparator): Patients received postoperative analgesia by intravenous fentanyl 10 µg/ml 3-8 mL/h.
  Interventions: Procedure: intravenous analgesia
- epiduaral infusion (Active Comparator): Patients received epidural analgesia intraoperatively with ropivacaine 0.75% 1 mg/kg and fentanyl 1 µg/kg followed by continuous epidural infusion of ropivacaine 0.2% 3-8 mL/h and fentanyl 2 µg/mL postoperatively.
  Interventions: Procedure: epidural infusion
- patient-controlled epidural analgesia (Active Comparator): In addition to epidural anesthesia and epidural infusion, postoperatively patients received patient-controlled epidural analgesia with ropivacaine/fentanyl bolus 1 mL, lock-out interval 12 min.
  Interventions: Procedure: patient-controlled epidural analgesia

INTERVENTIONS:
Procedure: intravenous analgesia — Patients received postoperative analgesia with intravenous infusion of fentanyl 10 µg/ml 3-8 mL/h
  Arms: intravenous analgesia
Procedure: epidural infusion — Postoperative analgesia was performed using continuous epidural infusion of ropivacaine 0.2% 3-8 mL/h and fentanyl 2 µg/mL
  Arms: epiduaral infusion
Procedure: patient-controlled epidural analgesia — Postoperative analgesia was performed by continuous epidural infusion of ropivacaine/fentanyl mixture combined with patient-controlled epidural analgesia with ropivacaine/fentanyl bolus 1 mL, lock-out interval 12 min.
  Arms: patient-controlled epidural analgesia

SUMMARY:
The aim of the present study was to assess the efficacy of thoracic epidural anesthesia followed by postoperative epidural infusion and patient-controlled epidural analgesia with ropivacaine/fentanyl in off-pump coronary artery bypass grafting

DETAILED DESCRIPTION:
Ninety-three patients were scheduled for off-pump coronary artery bypass (OPCAB) under propofol/fentanyl anesthesia. Day before surgery patients were asked for informed consent and randomized into three postoperative analgesia regimens aiming at a visual analog scale (VAS) score <30 mm at rest. The control group (n=31) received intravenous fentanyl 10 µg/ml postoperatively 3-8 mL/h. After placement of an epidural catheter at the level of Th2-Th4 before OPCAB, a thoracic epidural infusion (EI) group (n=31) received epidural anesthesia (EA) intraoperatively with ropivacaine 0.75% 1 mg/kg and fentanyl 1 µg/kg followed by continuous EI of ropivacaine 0.2% 3-8 mL/h and fentanyl 2 µg/mL postoperatively. The patient-controlled epidural analgesia (PCEA) group (n=31), in addition to EA and EI, received PCEA (ropivacaine/fentanyl bolus 1 mL, lock-out interval 12 min) postoperatively. Hemodynamics and blood gases were measured throughout 24 h after OPCAB.

ELIGIBILITY:
Inclusion Criteria:

* presence of coronary artery disease
* ASA II-III
* elective off-pump coronary artery bypass

Exclusion Criteria:

* age < 18 years
* severe valve dysfunction or peripheral vascular disease
* simultaneous interventions (carotid endarterectomy, aneurysm repair, etc.)
* transfer to CPB during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative mechanical ventilation | Participants will be followed for the duration of mechanical ventilation, an expected average of 6 hours
  Duration of postoperative mechanical ventilation, hours

SECONDARY OUTCOMES:
Hemodynamic stability | All period of operation and during 24 hours postoperatively
  Hemodynamic stability as assessed by mean arterial pressure, heart rate, cardiac index, requirement of inotrops/vasoactives and colloids

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y Kirov, Study Director — Northern State Medical University
Locations (1):
- Dep. of Anesthesiology, Northern SMU, Arkhangelsk, Russia

REFERENCES:
- [Derived] Kirov MY, Eremeev AV, Smetkin AA, Bjertnaes LJ. Epidural anesthesia and postoperative analgesia with ropivacaine and fentanyl in off-pump coronary artery bypass grafting: a randomized, controlled study. BMC Anesthesiol. 2011 Sep 18;11:17. doi: 10.1186/1471-2253-11-17. PMID 21923942